CLINICAL TRIAL: NCT00708929
Title: Does Complement Factor H Gene Polymorphism Play a Role in the Regulation of Vascular Tone in the Choroid?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Ass.Prof.Priv.Doz.Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-040607
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Genetic Polymorphism; Macular Degeneration; Regional Blood Flow; Ocular Physiology
Keywords: Age-related macular degeneration; Complement factor H; Choroidal blood flow
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): 14 subjects homozygous HH for the Tyr402His single nucleotide polymorphism
  Interventions: Procedure: Squatting
- 2 (Other): 14 subjects homozygous TT for the Tyr402His single nucleotide polymorphism
  Interventions: Procedure: Squatting

INTERVENTIONS:
Procedure: Squatting — Squatting for 6 minutes

SUMMARY:
Age related macular degeneration (AMD) is a multifactorial disease with a strong genetic component. Most importantly a genetic polymorphism in the gene encoding for the complement factor H (CFH) has been recently identified which is highly associated with an increased risk of developing AMD. This Tyr402His polymorphism located on chromosome 1q31 has been implicated to play a role in the development of the disease.

Given that it is known that impaired regulation of choroidal vascular tone is present in patients with AMD, the current study seeks to investigate whether the Tyr402His polymorphism is associated with altered choroidal autoregulation in healthy subjects. For this purpose a total of 100 healthy volunteers will be included in order to test the hypothesis that an impaired regulation of choroidal blood flow is present in subjects with homozygous Tyr402His variant.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years
* Nonsmokers
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropy less than 3 diopters

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Choroidal blood flow during isometric exercise | 10 minutes
Tyr402His genotyping | screening

SECONDARY OUTCOMES:
Mean arterial pressure | 20 minutes
Intraocular pressure | before and after blood flow measurements
Systolic/diastolic blood pressure | 20 minutes
Pulse rate | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhöfer, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria